CLINICAL TRIAL: NCT02140827
Title: Communication Through Instant Messaging Program for the Improvement of Bowel Preparation: a Two Centers Study
Brief Title: Instant Messaging Program (Wechat) Improve the Quality of Bowel Preparation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Air Force Military Medical University, China (Other)
Responsible Party: Principal Investigator, Yanglin Pan, Associated professor, Air Force Military Medical University, China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 20140508-5; 20140508-5 (Other: Ethics committee of Xijing Hospital)
Record Dates: First submitted 2014-05-14; First posted 2014-05-16 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Bowel Preparation
Keywords: bowel preparation; instant messaging program

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IMP education (Experimental): patients in this group are educated about bowel preparation by instant messaging program and meanwhile a booklet was also sent to them.
  Interventions: Other: IMP interactive education
- normal education (No Intervention): patients in this group are educated about bowel preparation on the day of reservation by nurse for about 15 minutes and meanwhile a booklet was also sent to them.

INTERVENTIONS:
Other: IMP interactive education — The detail and FAQ (Frequently Asked Questions) of bowel preparation instructions is delivered by Wechat.
  Other Names: Wechat education
  Arms: IMP education

SUMMARY:
Colonoscopy is the gold standard in the diagnosis of colorectal disease. The success of colonoscopy depends on high-quality bowel preparation by patients. Inadequate bowel cleansing reduces the cecal intubation rate, and the polyp detection rate (PDR). It also increases costs, mostly due to repeated procedures. The quality of bowel cleansing has remained suboptimal even though numerous different products and regimens have been tested and compared in no fewer than six meta-analyses. Therefore, a completely different approach to improve bowel cleansing is welcome.

Here the investigators assume that instant messaging program (Wechat) delivery the detail and FAQ (Frequently Asked Questions) of bowel preparation instructions would improve the quality of the bowel preparation. The Wechat program has some advantages, 1. Wechat supports over 400 million users, nearly half of the mobile subscribers population in China; 2. Wechat provided a real time communications including voice messages, pictures and text exchange timely; 3.Compare with telephone, Wechat is economical of both time and money; 4. Compare with bowel preparation instructional software and litera or cartoon educational booklet, Wechat is more interactive and responsive.

ELIGIBILITY:
Inclusion Criteria:

* age 18-80
* PEG as purgatives;
* using we-chat software by patients or their relatives
* outpatients

Exclusion Criteria:

* history of colorectal surgery
* known severe colonic stricture or obstructing tumor
* known or suspected bowel obstruction or perforation
* pregnant or lactating women
* patients who cannot give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2014-05; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Adequate bowel preparation quality at the time of colonoscopy defined by Ottawa score<6 | up to 5 months
  Ottawa score：A)cleanliness of each part of the colon: 0=excellent 1=good 2=fair 3=poor 4=inadequate B)fluid in whole colon: small=0 moderate=1 large=2
  The bowel preparation was considered inadequate if (1) inadequate visualization on colonoscopy defined by Ottawa score≥6; (2) the colonoscopy was cancelled because of poor bowel preparation; (3) incompleted colonoscopy because of inadequate bowel preparation (the Ottawa score was rated as 14 when patients with failed colonoscopy because of inadequate bowel preparation).

SECONDARY OUTCOMES:
Polyp detection rate | up to 5 months
  The proportion of participants with at least one polyp in each group
Compliance rate to instruction | up to 5 months
  The proportion of participants compliance to the instructions of diet and bowel preparation in each group
Willingness undergo a repeated bowel preparation | up to 5 months
  The number of participants have a willingness to undergo a repeated bowel preparation if needed

CONTACTS AND LOCATIONS:
Overall Officials: Yanglin Pan, M.D., Principal Investigator — Air Force Military Medical University, China; Limei Wang, M.D., Principal Investigator — Department of gastroenterology, Shaanxi Second People's Hospital
Locations (3):
- China (3):
  - Department of gastroenterology, Chancheng Central Hospital of Foshan, Foshan, Guangdong
  - Department of gastroenterology, Shaanxi Second People's Hospital, Xi'an, Shaanxi
  - Xijing Hospital of Digestive Diseases, Xi'an, Shaanxi

REFERENCES:
- [Derived] Kang X, Zhao L, Leung F, Luo H, Wang L, Wu J, Guo X, Wang X, Zhang L, Hui N, Tao Q, Jia H, Liu Z, Chen Z, Liu J, Wu K, Fan D, Pan Y, Guo X. Delivery of Instructions via Mobile Social Media App Increases Quality of Bowel Preparation. Clin Gastroenterol Hepatol. 2016 Mar;14(3):429-435.e3. doi: 10.1016/j.cgh.2015.09.038. Epub 2015 Oct 20. PMID 26492848